CLINICAL TRIAL: NCT05242107
Title: Role of Omega-3 Supplementation on Lipid Profile and Serum Leptin Level in Neonates With Intrauterine Growth Restriction
Brief Title: Omega-3 on Lipid Profile and Serum Leptin Level n Neonates With Intrauterine Growth Restriction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mai Rabie El-Sheikh, Doctor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35199/9/22
Record Dates: First submitted 2022-02-07; First posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Lipid Profile; Neonates; Intrauterine Growth Restriction
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega-3 supplement group (Experimental): This group included 35 full term Intrauterine Growth Restriction( IUGR) neonates, who received omega-3 supplement (Docosa-hexa-enoic acid (DHA) 40 mg/kg/ day) after establishment of full feeding.
  Interventions: Dietary Supplement: Omega-3 supplement group
- Full feeding without receiving any supplementation group (Experimental): This group included 35 full term Growth Restriction( IUGR) neonates who were followed up to full feeding without receiving any supplementation.
  Interventions: Other: Full feeding without receiving any supplementation group

INTERVENTIONS:
Dietary Supplement: Omega-3 supplement group — 35 Neonates were given Omega 3 in a dose of 40mg/kg/day (8), after establishment of full-feeding and for 2 weeks duration. Omega-300 (Montana pharmaceutical industry) capsule was used which contains 1000mg Omega 3 fatty acids.
  Arms: Omega-3 supplement group
Other: Full feeding without receiving any supplementation group — 35 full term Growth Restriction( IUGR) neonates who were followed up to full feeding without receiving any supplementation.
  Arms: Full feeding without receiving any supplementation group

SUMMARY:
The aim of our study will demonstrate the effect of omega 3 supplementation on serum lipid profile level and leptin level in neonates with Intrauterine Growth Restriction( IUGR)

DETAILED DESCRIPTION:
Intrauterine growth restriction is a major cause of perinatal mortality and morbidity .

It is noted to affect approximately 5-15 % of pregnant women. Egypt has one of the highest incidences of Intrauterine Growth Restriction. The incidence of IUGR varies among countries, populations, races and increases with decreasing gestational age. 14 to 20 million infants have been affected with Intrauterine Growth Restriction cases in the developing countries annually.

A complex and dynamic interaction of maternal, placental and fetal environment is involved in ensuring normal fetal growth. An imbalance or lack of coordination in this complex system may lead to Intrauterine Growth Restriction. Intrauterine Growth Restriction( IUGR) results in significant perinatal and long-term complications, including increased neonatal mortality and morbidity and higher risk for developing metabolic syndrome later in life.

Physiological differences have been noted in growth restricted infants. Intrauterine amino acid disturbances similar to biochemical changes seen in postnatal protein deprived states have been detected. Protein metabolism defect and altered lipid metabolism also have been described.

Undernourishment in utero appears to be associated with persisting changes in the metabolic functions. Birth weight influences the lipoprotein profile and cholesteryl ester transfer protein, which promotes a proatherogenic lipoprotein profile in plasma by determining chemical, physical and biological properties of the respective lipoprotein particle in neonates.

Recent research suggests that several of major disease of later life, including coronary heart disease, hypertension & type II diabetes originate in impaired intrauterine growth and development. These diseases may be consequence of programming whereby a stimulus or insult at a critical, sensitive period of early life has a permanent effect on structure, physiology and metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Any full-term Intrauterine growth restriction (IUGR) neonate

Exclusion Criteria:

* Preterm neonates
* Who died before feeding was established
* Multiple congenital anomalies including GIT anomalies
* Congenital infection
* Cholestasis
* Infant of diabetic mother (IDM)

Ages: 1 Day to 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Level of serum leptin | 4 weeks from admission to neonatal intensive care unit
  Effect of omega 3 (Docosa-hexa-enoic acid (DHA) 40 mg/kg/ day)supplementation on level of serum leptin in neonates with Intrauterine growth restriction (IUGR).

SECONDARY OUTCOMES:
Level of serum lipid | 4 weeks from admission to neonatal intensive care unit
  Effect of omega 3 (Docosa-hexa-enoic acid (DHA) 40 mg/kg/ day) supplementation on level of serum lipid in neonates with Intrauterine growth restriction (IUGR).

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta university, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The study will be available upon a reasonable request from the corresponding author
Supporting Information: Study Protocol
Time Frame: one year after the end of the study

REFERENCES:
- [Derived] Elsheikh M, El Amrousy D, El-Mahdy H, Dawoud H, Harkan A, El-Barky A. Lipid profile after omega-3 supplementation in neonates with intrauterine growth retardation: a randomized controlled trial. Pediatr Res. 2023 Oct;94(4):1503-1509. doi: 10.1038/s41390-023-02632-z. Epub 2023 May 18. PMID 37202530